CLINICAL TRIAL: NCT05343286
Title: Biological & Fonctional Signatures for Muscle Failures, Aged People & Personalized Physical Activity : BioFaSt MAPPA
Brief Title: Biological & Fonctional Signatures for Muscle Failures, Aged People & Personalized Physical Activity
Acronym: BioFaSt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-PP-24
Record Dates: First submitted 2022-03-02; First posted 2022-04-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Elderly
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- APAP group: adapted and personalized physical activity (Experimental): 12 weeks of adapted and personalized physical activity
  Interventions: Procedure: blood sample; Other: physical assessement; Behavioral: psychometric assessment
- APA group: adapted physical activity (Active Comparator): 12 weeks of generic physical activity
  Interventions: Procedure: blood sample; Other: physical assessement; Behavioral: psychometric assessment
- Control group: no physical activity (Sham Comparator): no physical activity
  Interventions: Procedure: blood sample; Other: physical assessement; Behavioral: psychometric assessment

INTERVENTIONS:
Procedure: blood sample — blood sample before and after 12 weeks of physical activity
Other: physical assessement — physical assessement before and after 12 weeks of physical activity
  * Standardized geriatric assessment (physician visit)
  * ICOPE Monitor Assessment
  * Sit-to-stand Test
  * Quantified Gait Analysis (QAM)
  * Bone densitometer measurement of body composition
Behavioral: psychometric assessment — Psychometric questionnaires
  * Cognitive tests (MMSE)
  * The long questionnaire of personality traits: Big Five Inventory
  * Perceived health and subjective age
  * Age group identification
  * Attitudes towards aging: French version of the Attitudes Toward Own Aging scale
  * Physical self-perception: French version of the Physical Self-Perception Profile
  * MOTIVATION SCALE FOR PA FOR HEALTH PURPOSES: Motivation Scale for Physical Activity in a Health Context
  * Aging Stereotypes and Exercise Scale

SUMMARY:
Physical activity is one of the most effective therapeutic interventions for frailty, sarcopenia or dynapenia. The benefits of physical activity processes are already widely documented. Typically, researchers want to understand the average response to an intervention to determine its overall effectiveness. However, sports trainers have understood it for a long time, the response of an athlete or a patient to training is very variable and the standard deviations present in all the scientific studies on the subject confirm it. There is therefore inter-individual variation in the response to exercise, with some subjects showing much greater improvements than others. Thus, one can wonder if this "non-response" following training is specific to the training modality. The effects of physical exercise on the body depend mainly on its type, intensity and duration. Thus, from a practical point of view, the most important perspective is the prediction and, ultimately, the individual optimization of management through physical activity.

DETAILED DESCRIPTION:
Main objective: To determine the effects of personalized physical activity management on the biological signatures of muscle failure.

Secondary objectives:

* Propose a support system through adapted and individualized physical activity, based on physical, biological and psycho-social indicators
* Identify the biological signatures (metabolomics, epigenetic) of muscle failure in the elderly.

Phenotype responders and non-responders in training

900 seniors (300 per group) APAP group: adapted and personalized physical activity APA group: adapted physical activity Control group: no physical activity

Total duration of the study 5 years, duration of participation for a patient 3 months; inclusion period: 57 months

Improvement of muscle failure in its broad definition (Strength, power, speed and lean mass)

) General data: description of characteristics with frequencies and percentage for categorical variables and with mean and standard deviation for quantitative variables.

ii) Analysis of the primary endpoint: Machine Learning (or supervised classification) and signaling pathway prediction approaches for statistical analysis and data interpretation.

iii) Analysis of secondary judgment criteria: approaches in Machine Learning (or supervised classification) and signaling pathway prediction for statistical analysis and interpretation of data with comparison of quantitative variables by Pearson correlation and categorical variables by t or chi 2 test depending on the case.

Adapt and individualize physical activity support for healthy or frail elderly people

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 60 years
* Affiliated patient or beneficiary of a social security scheme
* Patient having signed a prior informed consent.

Exclusion criteria

* Neurocognitive disorder preventing the expression of informed consent
* Patients protected by law under guardianship or curatorship, or who cannot participate in a clinical study under Article L. 1121-16 of the French Public Health Code
* Presence of a physical or cognitive pathology preventing the performance of the adapted physical activity protocol over 3 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
muscle power | before and after 12 week of physical activity program
  muscle power (Watt/Kg) assessed with the isokinetic ergometer.

SECONDARY OUTCOMES:
Different metabolomic signature (The amino acid composition) between the groups (APA, APAP, no physical activity) | at day 0
  Change in the amino acid composition (metabolomic signature) at Day 0 between the groups
Change in the amino acid composition (metabolomic signature) after 3 month of physical activity | between Day 0 and Month 3
  Change in the amino acid composition (metabolomic signature) after 3 month of physical activity for the APA and APAP groups compared to the no physical activity group
ICOPE Monitor Assessment | before and after 12 week of physical activity program
  Score of frailty. (Implementation of the Integrated Care of Older People, ICOPmonitor, 8 item, higher score means worse outcome)
Sit-to-stand Test | before and after 12 week of physical activity program
  number of movement
Quantified Gait Analysis (QAM) | before and after 12 week of physical activity program
  Gait velocity in m.s-1
Bone densitometer measurement of body composition | before and after 12 week of physical activity program
  % of lean mass
Cognitive tests | before and after 12 week of physical activity program
  Score Mini-Mental State Examination (MMSE, 0-30, higher score mean worse outcome)
The long questionnaire of personality traits | before and after 12 week of physical activity program
  Score of Big Five Inventory, 0-44, higher score means worse outcome
Perceived health (Score of the scale) | before and after 12 week of physical activity program
  Score of the scale, 0-6, higher score means better outcome
Subjective age | before and after 12 week of physical activity program
  Subjective age in years
Age group identification (Years) | before and after 12 week of physical activity program
  Age group identification in years
Attitudes towards aging | before and after 12 week of physical activity program
  Score on the French version of the Attitudes Toward Own Aging scales, 0-7, higher score means better outcome
Physical self-perception | before and after 12 week of physical activity program
  Score on the French version of the Physical Self-Perception Profile, 0-6, higher score means better outcome
Motivation scale for physical activity for health purposes | before and after 12 week of physical activity program
  Score on the Motivation Scale for Physical Activity in a Health Context,0-30, higher score means better outcome
Aging Stereotypes and Exercise Scale | before and after 12 week of physical activity program
  Score on the French Aging Stereotypes and Exercise Scale (ASES), 0-12, higher score means better outcome
Improvement of muscle force | before and after 12 week of physical activity program
  Improvement of muscle force (N/Kg) assessed with the isokinetic ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, PU-PH, Principal Investigator — geriatric Department
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No